CLINICAL TRIAL: NCT05200936
Title: Safety and Efficacy of Repeated Low Dose d-Lysergic Acid Diethylamide (LSD) D-tartrate (MM-120) as Treatment for ADHD in Adults: a Multi-center, Randomized, Double-blind, Placebo-controlled Phase 2a Proof of Concept Trial
Brief Title: Safety and Efficacy of Low Dose MM-120 for ADHD Proof of Concept Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Definium Therapeutics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MMED007
Record Dates: First submitted 2021-12-21; First posted 2022-01-21 (Actual); Results first posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: ADHD; Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1- Placebo (Placebo Comparator): A total of 26 patients will receive a placebo identical in appearance to the investigational medicinal product (IMP) administered orally twice weekly (e.g., Tuesday/Friday) for 6 weeks.
  Interventions: Other: Placebo
- Arm 2- MM-120 (Experimental): A total of 26 patients will receive 20 μg of MM-120 administered orally twice weekly for 6 weeks.
  Interventions: Drug: MM-120

INTERVENTIONS:
Drug: MM-120 — MM-120 is a psychedelic drug that can cause intensified thoughts, emotions, and sensory perception. At sufficiently high dosages MM-120 manifests primarily visual, as well as auditory, hallucinations.
  Arms: Arm 2- MM-120
Other: Placebo — A treatment which is designed to have no therapeutic value.
  Arms: Arm 1- Placebo

SUMMARY:
This study measures the safety and efficacy of repeated low dose MM-120 as treatment for ADHD in adults: a multi-center, randomized, double-blind, placebo-controlled

DETAILED DESCRIPTION:
This study is a multi-center, randomized, double-blind, placebo-controlled Phase 2a study of low dose MM-120 (20 μg) compared with a placebo administered for 6 weeks (twice a week on a 3/4-day schedule).

Low dose MM-120 (20 μg) is about 20% of the dose typically consumed for recreational psychedelic purposes.

There will be a 1:1 randomization, double-blind, to MM-120 or placebo with the aim to reach 26 evaluable patients in each of the 2 arms at Week 6.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients ≥ 18 and ≤ 65 years of age at Screening
* Patients with the diagnosis of Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) ADHD, as determined by clinical evaluation and confirmed by structured interview (MINI).
* Adequate organ function.
* Able to understand the study procedures and understand risks associated with the study, and sign written informed consent to participate in the study.
* Must be willing to refrain from more than 6 standard alcoholic drinks a week, more than 10 cigarettes a day, and more than 2 cups of coffee a day throughout the study treatment period (6 weeks) and until the last study visit is complete.

Exclusion Criteria:

* Past or present diagnosis of a primary psychotic disorder or first degree relative with a psychotic disorder.
* Past or present bipolar disorder (DSM-5).
* Any lifetime history of suicide attempt.
* Once Informed Consent form is signed, not willing or able to stop any prescription or non-prescription ADHD medications.
* Use of investigational medication/treatment in the past 30 days.
* Patients with a positive urine drug screen with the exception of THC or its metabolites.
* Pregnant or nursing females.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Kuypers, Principal Investigator — Maastricht University; Matthias Liechti, Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Maastricht University, Maastricht, Netherlands
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller L, Santos de Jesus J, Schmid Y, Muller F, Becker A, Klaiber A, Straumann I, Luethi D, Haijen ECHM, Hurks PPM, Kuypers KPC, Liechti ME. Safety and Efficacy of Repeated Low-Dose LSD for ADHD Treatment in Adults: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Jun 1;82(6):555-562. doi: 10.1001/jamapsychiatry.2025.0044. PMID 40105807

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 74 potential participants were screened and 21 were excluded.
Period: Overall Study
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Started | 27 | 26
Completed | 23 | 23
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: A summary of demographic information for the FAS is shown below.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo | Total
Number analyzed (Participants) | 27 | 26 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (12.8) | 33.1 (11.0) | 36.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 14 | 17 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 27 | 26 | 53
Region of Enrollment [Number; unit: participants]
  Netherlands | 2 | 1 | 3
  Switzerland | 25 | 25 | 50
Baseline ADHD investigator symptom rating scale (AISRS) [Mean (Standard Deviation); unit: units on a scale] — The Adult ADHD investigator symptom rating scale (AISRS) total score consists of 18 items from the original Attention-deficit/hyperactivity Disorder Rating Scale (ADHD-RS). The ADHD-RS includes 9 items that address symptoms of inattention, and 9 items that address symptoms of impulsivity and hyperactivity. Each item is rated from 0 to 3. The AISRS total score can range from 0 to 54. A higher score corresponds to a worse severity of ADHD. Population: Baseline values from subjects not included in Primary efficacy analysis were excluded from this calculation
  units on a scale
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 37.4 (6.11) | 37.3 (5.24) | 37.4 (5.69)

OUTCOME MEASURES:

1. Primary Outcome: Change in Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Symptoms
Description: The Adult ADHD investigator symptom rating scale (AISRS) total score consists of 18 items from the original Attention-deficit/hyperactivity Disorder Rating Scale (ADHD-RS). The ADHD-RS includes 9 items that address symptoms of inattention, and 9 items that address symptoms of impulsivity and hyperactivity. Each item is rated from 0 to 3. The AISRS total score can range from 0 to 54. A higher score corresponds to a worse severity of ADHD.
Time Frame: 6 weeks
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 23 | 23
units on a scale
  Baseline | 37.4 (6.11) | 37.3 (5.24)
  Week 6 | 29.6 (8.27) | 29.0 (8.47)
Statistical Analysis 1: Comparison: Arm 2- MM-120 vs Arm 1- Placebo; Test type: Superiority; p = 0.7145, Mixed Models Analysis — p-value is 1-sided

2. Secondary Outcome: Changes in Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Investigator Symptom Rating Scale (AISRS) Symptoms
Description: as for outcome 1
Time Frame: Week 2
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 26 | 26
units on a scale
  Baseline | 37.5 (5.76) | 36.9 (5.10)
  Week 2 | 34.2 (6.49) | 32.1 (4.96)
Statistical Analysis 1: Comparison: Arm 2- MM-120 vs Arm 1- Placebo; Test type: Superiority; p = 0.9613, ANCOVA

3. Secondary Outcome: Number of Patients Who Experience a Decrease in the Clinical Global Impressions Scale (CGI-S)
Description: The Clinical Global Impression - Severity (CGI-S) was used to assess the subject's current severity of illness at the time of the assessment relative to the clinician's past experience with patients who have the same diagnosis. The CGI-S comprises 1 Investigator-completed (or trained rater-completed) item with 7 possible ratings (1-7 points), where a higher score indicates more severe illness.
Time Frame: Baseline, Week 2, Week 6, Week 10
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 27 | 26
Participants
  Baseline to Week 2 | 8 | 11
  Baseline to Week 6 | 16 | 15
  Baseline to Week 10 | 17 | 12

4. Secondary Outcome: Change From Baseline in in Clinical Global Impressions Scale (CGI-S)
Description: as for outcome 3
Time Frame: Baseline, Week 2, Week 6
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 27 | 26
units on a scale
  Baseline for Week 2: number analyzed (Participants) | 26 | 26
  Baseline for Week 2 | 4.9 (0.71) | 4.7 (0.62)
  Week 2: number analyzed (Participants) | 26 | 26
  Week 2 | 4.6 (0.70) | 4.3 (0.53)
  Baseline for Week 6: number analyzed (Participants) | 23 | 23
  Baseline for Week 6 | 4.9 (0.73) | 4.8 (0.60)
  Week 6: number analyzed (Participants) | 23 | 23
  Week 6 | 4.0 (0.88) | 3.8 (0.85)

5. Secondary Outcome: Adult Attention-deficit/Hyperactivity Disorder Self-reporting Rating Scale (ASRS)
Description: The Adult Attention-Deficit/Hyperactivity Disorder Self-Reporting Rating Scale (ASRS) is composed of 18 questions, and uses a scale that ranges from 0-4 based on the individuals mark in either the "never, rarely, sometimes, often, very often" column for a possible total score of 72. A higher score corresponds to a worse severity of ADHD.
Time Frame: 6 weeks
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 27 | 26
units on a scale
  Baseline for Week 2: number analyzed (Participants) | 25 | 26
  Baseline for Week 2 | 48.0 (7.01) | 43.9 (7.33)
  Week 2: number analyzed (Participants) | 25 | 26
  Week 2 | 40.2 (9.26) | 36.7 (9.38)
  Baseline for Week 4: number analyzed (Participants) | 17 | 18
  Baseline for Week 4 | 48.6 (7.67) | 44.6 (7.61)
  Week 4: number analyzed (Participants) | 17 | 18
  Week 4 | 35.2 (8.14) | 34.9 (9.29)
  Baseline for Week 6 (Day 36): number analyzed (Participants) | 20 | 23
  Baseline for Week 6 (Day 36) | 48.4 (7.10) | 44.2 (7.72)
  Week 6 (Day 36): number analyzed (Participants) | 20 | 23
  Week 6 (Day 36) | 36.0 (9.99) | 33.1 (11.70)
  Baseline to Week 6 (Day 40): number analyzed (Participants) | 17 | 22
  Baseline to Week 6 (Day 40) | 49.6 (6.96) | 44.0 (7.86)
  Week 6 (Day 40): number analyzed (Participants) | 17 | 22
  Week 6 (Day 40) | 31.0 (9.18) | 31.7 (12.0)

6. Secondary Outcome: Change From Baseline in Connors' Adult ADHD Rating Scale (CAARS)
Description: The Connors' Adult ADHD Rating Scale (CAARS) Self-Report Long Form is a 66-item measure of ADHD symptom. Responses are scored on a 4-point scale, where 0 = not at all, 1 = just a little, 2 = pretty much, and 3 = very much. Item scores are summed to three main scores which are then transformed using population-derived age- and sex-adjusted norm values to a T-score. A T-score < 60 indicates no ADHD. A T-score of 60-64 indicates borderline ADHD. A T-score of > 64 indicates ADHD.
Time Frame: 6 weeks
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 27 | 26
units on a scale
  Change from baseline to Week 2: number analyzed (Participants) | 26 | 26
  Change from baseline to Week 2 | -4.0 (5.79) | -2 (3.29)
  Change from baseline to Week 4: number analyzed (Participants) | 18 | 18
  Change from baseline to Week 4 | -6.9 (5.36) | -3.6 (4.4)
  Change from Baseline to Week 6 (Day 36): number analyzed (Participants) | 21 | 23
  Change from Baseline to Week 6 (Day 36) | -5.6 (6) | -4.6 (5.1)
  Change from Baseline to Week 6 (Day 40): number analyzed (Participants) | 18 | 21
  Change from Baseline to Week 6 (Day 40) | -6.3 (5.82) | -4.3 (5.98)

7. Secondary Outcome: 5 Dimensions of Altered States of Consciousness Questionnaire (5D-ASC) Scores
Description: The 5 dimensions of altered states of consciousness (5D-ASC) scale is a visual analog scale (VAS) consisting of 94 items each scored on a 0-100mm VAS extrapolated to 100% scale for quantitative evaluation. These 94 items are categorized into five dimensions: oceanic boundlessness (min:0, max:2700), anxious ego dissolution (min:0, max:2100), visionary destructuralization (min:0, max:1800), auditory alterations (min:0, max:1600), and vigilance reduction (min:0, max:1200). The total score is the sum of all questions and can range from 0 to 9400. Higher scores = more alteration in state of consciousness.
Time Frame: 6 weeks
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 27 | 26
units on a scale
  W1D1 Oceanic boundlessness | 479.6 [277.3 to 681.9] | 161.3 [26.2 to 296.4]
  W1D1 Anxious ego dissolution | 103.6 [35.5 to 171.6] | 19.0 [5.9 to 32.2]
  W1D1 Visionary destructuralization | 233.4 [135.6 to 331.2] | 94.8 [18.6 to 171.0]
  W1D1 Auditory alterations | 71.0 [12.2 to 129.7] | 32.7 [1.6 to 63.8]
  W1D1 Vigilance reduction | 288.5 [198.0 to 379.0] | 155.2 [79.3 to 231.1]
  W1D1 Total score | 1176.0 [781.4 to 1570.6] | 463.0 [166.9 to 759.1]
  W6 Oceanic boundlessness: number analyzed (Participants) | 23 | 23
  W6 Oceanic boundlessness | 403.3 [194.3 to 612.4] | 70.2 [16.0 to 124.4]
  W6 Anxious ego dissolution: number analyzed (Participants) | 23 | 23
  W6 Anxious ego dissolution | 41.0 [-0.6 to 82.7] | 4.2 [-0.4 to 8.7]
  W6 Visionary destructuralization: number analyzed (Participants) | 23 | 23
  W6 Visionary destructuralization | 199.7 [86.9 to 312.5] | 32.9 [6.4 to 59.4]
  W6 Auditory alterations: number analyzed (Participants) | 23 | 23
  W6 Auditory alterations | 18.4 [0.2 to 36.7] | 4.2 [0.0 to 8.4]
  W6 Vigilance reduction: number analyzed (Participants) | 23 | 23
  W6 Vigilance reduction | 90.3 [52.2 to 128.5] | 20.0 [6.9 to 33.1]
  W6 Total scores: number analyzed (Participants) | 23 | 23
  W6 Total scores | 752.9 [387.2 to 1118.6] | 131.4 [50.0 to 212.8]

8. Secondary Outcome: Mystical Experience Questionnaire 30 Items (MEQ30)
Description: The Mystical Experience Questionnaire 30 item (MEQ30) is a 30-item questionnaire rated on a six-point scale. The scale has been used to assess mystical experiences in studies using psilocybin and LSD. Higher scores = greater mystical experiences. The total score is expressed as a percentage of the maximum possible score (0 to 100%).
Time Frame: 6 weeks
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized.
Measure: Mean (95% Confidence Interval); unit: percentage of maximum possible score
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 27 | 26
percentage of maximum possible score
  Week 1 Day 1 | 22.37 [14.57 to 30.17] | 10.40 [3.97 to 16.84]
  Week 6: number analyzed (Participants) | 23 | 22
  Week 6 | 20.50 [11.94 to 29.06] | 5.20 [1.40 to 9.01]

9. Secondary Outcome: Summary of Drug Effects Visual Analog Scale (VAS)
Description: A series of single item visual Analog Scales (VAS) are used repeatedly 0 -6 hours after drug administration: The following 9 items were used in VAS (0-100 mm): "any drug effect", "good drug effect", bad drug effect", "drug liking", "fear", nausea", "alteration of vision", "alteration of sense of time", and "the boundaries between myself and my surroundings seem to blur". VAS scores range from 0 = no effect to 100 = strong effect. The scores for each item are extrapolated to a 100% scale and presented for each time point of assessment.
Time Frame: 6 hours
Population: Full Analysis Set (FAS): All subjects in the randomized set (RAN) who were not mis-randomized.
Measure: Mean (Full Range); unit: percentage of maximum possible score
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
Number analyzed (Participants) | 27 | 26
percentage of maximum possible score
  0h Any drug effect | 0 [0 to 0] | 0 [0 to 0]
  0h Drug liking | 37.1 [0 to 55] | 44.9 [0 to 52]
  0h Fear | 2.7 [0 to 36] | 1.4 [0 to 23]
  0h Nausea | 1.1 [0 to 30] | 0 [0 to 0]
  0h Alteration of vision | 0 [0 to 0] | 0 [0 to 0]
  0h Alteration of sense of time | 0 [0 to 0] | 0 [0 to 0]
  0h Boundaries blur | 0 [0 to 0] | 0 [0 to 0]
  0.5h Any drug effect | 8.9 [0 to 78] | 11.3 [0 to 75]
  0.5h Drug liking | 44.4 [0 to 78] | 48.1 [0 to 83]
  0.5h Fear | 2.0 [0 to 54] | 2.2 [0 to 48]
  0.5h Nausea | 2.0 [0 to 53] | 0.2 [0 to 3]
  0.5h Alteration of vision | 3.5 [0 to 54] | 7.4 [0 to 81]
  0.5h Alteration of sense of time | 2.5 [0 to 41] | 3.2 [0 to 35]
  0.5h Boundaries blur | 3.0 [0 to 71] | 0.8 [0 to 12]
  1h Any drug effect | 24.1 [0 to 100] | 12.7 [0 to 64]
  1h Drug liking | 49.7 [0 to 97] | 51.8 [2 to 97]
  1h Fear | 1.4 [0 to 32] | 0.1 [0 to 2]
  1h Nausea | 2.7 [0 to 37] | 1.0 [0 to 23]
  1h Alteration of vision | 4.0 [0 to 56] | 6.9 [0 to 72]
  1h Alteration of sense of time | 8.1 [0 to 73] | 6.3 [0 to 68]
  1h Boundaries blur | 6.0 [0 to 87] | 1.5 [0 to 24]
  2h Any drug effect | 38.1 [0 to 97] | 12.8 [0 to 72]
  2h Drug liking | 57.3 [0 to 100] | 53.3 [3 to 100]
  2h Fear | 4.1 [0 to 68] | 0.1 [0 to 2]
  2h Nausea | 8.2 [0 to 60] | 0.1 [0 to 2]
  2h Alteration of vision | 13.0 [0 to 84] | 6.2 [0 to 88]
  2h Alteration of sense of time | 13.5 [0 to 78] | 4.4 [0 to 53]
  2h Boundaries blur | 12.3 [0 to 83] | 1.3 [0 to 14]
  3h Any drug effect | 44.3 [0 to 97] | 11.1 [0 to 65]
  3h Drug liking | 61.6 [0 to 100] | 53.1 [3 to 96]
  3h Fear | 2.9 [0 to 54] | 0.2 [0 to 2]
  3h Nausea | 8.0 [0 to 56] | 0.2 [0 to 3]
  3h Alteration of vision | 13.9 [0 to 84] | 6.5 [0 to 76]
  3h Alteration of sense of time | 12.3 [0 to 89] | 4.9 [0 to 74]
  3h Boundaries blur | 12.7 [0 to 88] | 1.4 [0 to 31]
  4h Any drug effect | 38.5 [0 to 97] | 15.1 [0 to 100]
  4h Drug liking | 60.7 [0 to 100] | 48.0 [2 to 100]
  4h Fear | 2.7 [0 to 50] | 0.1 [0 to 2]
  4h Nausea | 6.9 [0 to 65] | 0.1 [0 to 2]
  4h Alteration of vision | 12.4 [0 to 86] | 3.2 [0 to 37]
  4h Alteration of sense of time | 12.1 [0 to 92] | 7.0 [0 to 57]
  4h Boundaries blur | 6.9 [0 to 69] | 0.2 [0 to 2]
  6h Any drug effect | 16.7 [0 to 75] | 9.6 [0 to 72]
  6h Drug liking | 54.8 [0 to 100] | 49.6 [0 to 100]
  6h Fear | 2.3 [0 to 52] | 2.1 [0 to 48]
  6h Nausea | 3.6 [0 to 52] | 0.2 [0 to 4]
  6h Alteration of vision | 4.1 [0 to 59] | 5.8 [0 to 59]
  6h Alteration of sense of time | 6.3 [0 to 69] | 3.0 [0 to 55]
  6h Boundaries blur | 4.1 [0 to 61] | 0.1 [0 to 2]

10. Other Pre Specified Outcome: Pharmacokinetic Outcomes
Description: Maximum Plasma Concentration [Cmax] of MM-120 in the blood at Week 1 Day 1
Time Frame: 0.5, 1, 2, 3, 4, 6 hours post-dose
Population: Pharmacokinetic Set (PKS): All subjects in the randomized set (RAN) who received a dose of MM120 and had at least 1 postdose PK measurement without important protocol deviations thought to significantly affect the PK of the drug. A strategy for dealing with data affected by protocol violations and deviations was to be agreed to by the Sponsor, monitor, and pharmacokineticist, prior to clean file and code break. Subjects were analyzed according to the treatment they actually received.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 2- MM-120
Number analyzed (Participants) | 24
ng/mL
  Pre-dose (0 hours) | 0 (0)
  0.5hours | 0.3250 (0.16534)
  1hour | 0.4410 (0.15686)
  2hours | 0.4270 (0.12832)
  3hours | 0.3591 (0.12493)
  4hours | 0.3066 (0.10851)
  6hours | 0.2117 (0.09361)

11. Other Pre Specified Outcome: Pharmacokinetic Parameters (Cmax)
Description: Maximum concentration (Cmax)
Time Frame: 0.5, 1, 2, 3, 4, 6 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 2- MM-120
Number analyzed (Participants) | 24
ng/mL | 0.4811 (0.14279)

12. Other Pre Specified Outcome: Pharmacokinetic Parameters (Tmax and t1/2)
Description: Time to maximum concentration (Tmax), half life (t1/2)
Time Frame: 0.5, 1, 2, 3, 4, 6 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm 2- MM-120
Number analyzed (Participants) | 24
hours
  Tmax | 1.46 (0.706)
  t1/2 | 3.8187 (1.27269)

13. Other Pre Specified Outcome: Pharmacokinetic Parameters (AUC0-inf and AUC0-6h)
Description: Area under the concentration curve from time 0 to infinity (AUC0-inf), Area under the concentration curve from time 0 to 6 hour (AUC0-6h)
Time Frame: 0.5, 1, 2, 3, 4, 6 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Arm 2- MM-120
Number analyzed (Participants) | 24
ng*h/mL
  AUC0-inf | 3.2450 (1.58494)
  AUC0-6hr | 1.9411 (0.63490)

ADVERSE EVENTS:
Time Frame: From time of signing ICF (or screening visit) through study completion, typically 14 weeks.
Description: Each event was to be described in detail, along with start and stop dates, severity, relationship to IMP, action taken, and outcome. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) as specified in the SAP.
Arm/Group | Arm 2- MM-120 | Arm 1- Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 21/27 | 23/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 2- MM-120 (N=27) | Arm 1- Placebo (N=26)
Headache (Nervous system disorders) | 13 | 9
Disturbance in Attention (Nervous system disorders) | 2 | 2
Akathisia (Nervous system disorders) | 1 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Restless leg syndrome (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Illusion (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Apathy (Psychiatric disorders) | 1 | 2
Euphoric mood (Psychiatric disorders) | 1 | 0
Flashbacks (Psychiatric disorders) | 1 | 0
Hypersomnia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 4 | 1
Feeling abnormal (General disorders) | 2 | 0
Swelling (General disorders) | 1 | 0
Full blood count abnormal (Investigations) | 1 | 0
Heart rate increased (Investigations) | 0 | 1
Pregnancy test positive (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Urine cannabinoids increased (Investigations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Palate injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Syncope (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hot flush (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Urethritis noninfective (Renal and urinary disorders) | 0 | 1
Premenstrual pain (Reproductive system and breast disorders) | 0 | 1
High risk sexual behaviour (Social circumstances) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
Although a multicenter-trial, one site enrolled 95% of participants. Only twice-weekly dose regimen was tested, which may not account for interindividual variability in response. Finally, other outcomes such as emotion regulation were not addressed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Sponsor has at least 30-60 days to review a proposed publication before submission for purposes of requesting the removal of Sponsor's confidential information.
2. PI's will not publish or disclosure their single-site data prior to a multi-center publication of the aggregate study data, unless Sponsor does not publish a multi-center publication within 12 months following conclusion of the overall study.

DOCUMENTS (2):
  • Study Protocol (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT05200936/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT05200936/SAP_001.pdf